CLINICAL TRIAL: NCT02023866
Title: An Open-Label, Dose-Escalating Study to Assess the Safety, Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamics of Cysteamine Bitartrate Delayed-release Capsules (RP103) for Treatment of Children With Inherited Mitochondrial Disease
Brief Title: Open-Label, Dose-Escalating Study Assessing Safety, Tolerability, Efficacy, of RP103 in Mitochondrial Disease
Acronym: MITO-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP103-MITO-001
Record Dates: First submitted 2013-12-17; First posted 2013-12-30 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Inherited Mitochondrial Disease, Including Leigh Syndrome
Keywords: Leigh Syndrome; Leber's hereditary optic neuropathy; myoclonic epilepsy; mitochondrial encephalomyopathy; Kearn-Sayre syndrome; POLG-related disorders; Neurogastrointestinal encephalopathy
MeSH Terms: conditions — Leigh Disease; Optic Atrophy, Hereditary, Leber; Epilepsies, Myoclonic; Mitochondrial Encephalomyopathies; Ophthalmoplegia, Chronic Progressive External | interventions — Cysteamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cysteamine Bitartrate Delayed-release (Experimental): Cysteamine bitartrate delayed-release capsules were administered twice daily following a dose-escalation design with a progressive weekly dose increase over the first 6 weeks. The starting dose was 0.2 g/m²/day, up to a maximum dose of 1.3 g/m²/day. Participants remained on their highest tolerated dose until Week 24.
  Interventions: Drug: Cysteamine Bitartrate

INTERVENTIONS:
Drug: Cysteamine Bitartrate — Cysteamine Bitartrate Delayed-release capsules
  Other Names: RP103

SUMMARY:
To evaluate safety, tolerability and efficacy of cysteamine bitartrate delayed-release capsules (RP103) administered at a target maintenance dose of 1.3 g/m²/day in two divided doses, every 12 hours, for up to 6 months in patients with inherited mitochondrial disease.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation study to assess the safety, tolerability, efficacy, pharmacokinetics and pharmacodynamics of cysteamine bitartrate delayed-release capsules (RP103) for treatment of children with inherited mitochondrial disease.

Prior to treatment, patients will undergo a Screening Visit. If eligible, each participant will return for the Day 1 study visit and begin dosing. Every 2 weeks over the subsequent 8 weeks, participants will alternate between returning to the clinic for detailed assessments (Weeks 4 and 8) and receiving a telephone call from the Investigator team to assess safety and RP103 dose (Weeks 2 and 6) and the potential need for an immediate unscheduled study visit. Thereafter, participants will continue to return to the clinic every 4 weeks for detailed assessments at Weeks 12, 16, 20, and 24 (the Study Exit visit).

The Study Exit visit will occur at Week 24, and participants will be offered the opportunity to continue on to an extension study (RP103-MITO-002 [NCT02473445]) until results of the present study are known.

Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 6 years and < 18 years
2. Body weight ≥ 5 kg
3. Documented (genetically confirmed known mutation, i.e. no variants of uncertain significance) diagnosis of inherited mitochondrial disease other than Friedreich's ataxia (FRDA)
4. Moderate disease severity based on Newcastle Pediatric Mitochondrial Disease Scale (NPMDS) score, with a score between 15 to 45 inclusive [Leber's Hereditary Optic Neuropathy (LHON) subjects are exempt of this inclusion criteria], if approved by the sponsor.
5. For patients regularly taking dietary supplements such as creatinine, alpha-lipoic acid, coenzyme Q10 (CoQ10), vitamin B, carnitine, etc. they have to have been taking them for at least 3 months pre-study and will agree to keep these the same throughout the study (from the Screening Visit to Study Exit)
6. With respect to concomitant medications, the subject must:

   1. Be willing to abstain from initiating dietary supplements and non-prescribed medications, except as allowed by the Investigator, throughout the study (from the Screening Visit to Study Exit);
   2. Be on a stable dose of medications prescribed for seizure management and prevention. Stable dose in this context means unchanged for at least 30 days prior to the Screening Visit.
7. Willing and able to comply with study drug dosing requirements, i.e. ingest the RP103 capsules intact, or sprinkled in liquid or soft food, or using a g-tube
8. Sexually active female subjects of childbearing potential (i.e., not surgically sterile [tubal ligation, hysterectomy, or bilateral oophorectomy]) must agree to utilize two of the following acceptable forms of contraception throughout the study (from the Screening Visit to Study Exit):

   1. Hormonal contraception: birth control pills, injection, patch, vaginal ring or implant;
   2. Condom or diaphragm, with spermicide;
   3. Intrauterine device (IUD)
   4. Sterile male partner (vasectomy performed at least 6 months prior to the study).
9. Subjects's legally authorized representative must provide written informed consent; Subject must provide assent, if required by local/institutional requirements
10. Have mitochondrial myopathy as evidenced by one or more of the following criteria:

    1. Weakness consistent with myopathy (e.g. accompanied by muscle wasting and/or absence of neuropathy) on physical exam
    2. OR documented myopathy on the basis of muscle biopsy consistent with mitochondrial myopathy disease
    3. OR weakness and/or progressive exercise intolerance (in which modest exercise typically provokes heaviness, weakness, aching of active muscles, or tachycardia). Weakness should be due to myopathy and not neuropathy or other causes as deemed by investigator

Exclusion Criteria:

1. Documented diagnosis of concurrent inborn errors of metabolism
2. Non-elective hospitalization related to mitochondrial disease or direct complication of disease within 60 days prior to the Screening Visit.
3. Platelet count, lymphocyte count or hemoglobin below the lower limit of normal (LLN) at the Screening Visit
4. Hepatic insufficiency with liver enzyme tests (alkaline phosphatase, aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) greater than 2.5 times the upper limit of normal (ULN) at the Screening Visit
5. Bilirubin > 1.2 g/dL at the Screening Visit
6. Inability to complete the elements of the study, e.g., coma, hemodynamic instability or requiring continuous ventilator support.
7. Malabsorption requiring total parenteral nutrition (TPN), chronic diarrhea, bouts of pseudo obstruction
8. Severe end-organ hypo-perfusion syndrome secondary to cardiac failure resulting in lactic acidosis
9. Patients with suspected elevated intracranial pressure, pseudotumor cerebri (PTC) and/or papilledema
10. Severe gastrointestinal disease including gastroparesis
11. History of angina, myocardial infarction, or cardiac surgery within 2 years prior to the Screening Visit
12. Any clinically significant electrocardiogram (ECG), including dysrhythmia, or clinically significant abnormal laboratory finding not already listed above at the Screening Visit
13. History of drug or alcohol abuse
14. History of pancreatitis
15. Participated in an investigational drug trial within 30 days or, within 90 days for a biologic, device, or surgical treatment, for inherited mitochondrial diseases prior to the Screening Visit
16. Known or suspected hypersensitivity to cysteamine and penicillamine
17. Female subjects who are nursing, planning a pregnancy, known or suspected to be pregnant, or with a positive serum pregnancy test at the Screening Visit
18. Subject's who, in the opinion of the Investigator, are not able or willing to comply with the protocol.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- United States (5):
  - University of California at San Diego (UCSD), San Diego, California
  - Stanford University, Stanford, California
  - Akron Children's Hospital, Akron, Ohio
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Division of Medical Genetics, Salt Lake City, Utah

REFERENCES:
- [Background] Bousquet M, Gibrat C, Ouellet M, Rouillard C, Calon F, Cicchetti F. Cystamine metabolism and brain transport properties: clinical implications for neurodegenerative diseases. J Neurochem. 2010 Sep;114(6):1651-8. doi: 10.1111/j.1471-4159.2010.06874.x. Epub 2010 Aug 19. PMID 20569301
- [Background] Salmi H, Leonard JV, Rahman S, Lapatto R. Plasma thiol status is altered in children with mitochondrial diseases. Scand J Clin Lab Invest. 2012 Apr;72(2):152-7. doi: 10.3109/00365513.2011.646299. Epub 2012 Jan 2. PMID 22208644
- [Background] Maher P, Lewerenz J, Lozano C, Torres JL. A novel approach to enhancing cellular glutathione levels. J Neurochem. 2008 Nov;107(3):690-700. doi: 10.1111/j.1471-4159.2008.05620.x. Epub 2008 Aug 12. PMID 18702664
- [Background] Mancuso M, Orsucci D, Logerfo A, Rocchi A, Petrozzi L, Nesti C, Galetta F, Santoro G, Murri L, Siciliano G. Oxidative stress biomarkers in mitochondrial myopathies, basally and after cysteine donor supplementation. J Neurol. 2010 May;257(5):774-81. doi: 10.1007/s00415-009-5409-7. Epub 2009 Dec 4. PMID 19960200

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cysteamine Bitartrate Delayed-release
Started | 36
Completed | 30
Not Completed | 6
Not completed — Non-compliance | 2
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Black of African American | 0
  Native Hawaiian or other Pacific Islander | 0
  White | 28
  Other | 2
  Multiple | 3
Mitochondrial Disease Subtype [Count of Participants; unit: Participants] — LHON = leber hereditary optic neuropathy; MELAS = mitochondrial encephalomyopathy, lactic acidosis, and strokelike syndrome MERFF = myoclonic epilepsy and ragged-red fibers; NUBPL = Nucleotide Binding Protein-Like; POLG = Polymerase (DNA Directed), Gamma.
  Participants
    Leigh Syndrome | 9
    POLG-related disorders | 7
    MELAS | 6
    MERFF | 4
    Others | 4
    LHON | 3
    NUBPL Related Encephalopathy | 2
    Kearns-Sayre syndrome | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Newcastle Paediatric Mitochondrial Disease Scale (NPMDS) Sections I-IV
Description: The NPMDS evaluates the progression of mitochondrial disease in pediatric patients in 4 domains:
  I - Current Function (vision, hearing, communication, feeding, and mobility) with scores ranging from 0 to 21; II -System Specific Involvement (seizures, encephalopathy, bleeding diathesis or coagulation defects, gastrointestinal, endocrine, respiratory, cardiovascular, renal, liver, and blood) with scores ranging from 0 to 30.
  III - Current Clinical Assessment (growth and development over past 6 months, vision, strabismus and eye movement, myopathy, ataxia, pyramidal, extrapyramidal, and neuropathy) with scores ranging from 0 to 28; and IV - Quality of Life with scores ranging from 0 to 25. For sections I-III, higher scores reflect more severe disease. For Section IV, a higher score reflects a lower quality of life.
Time Frame: Baseline through Week 24
Population: Completers Analysis Set included all participants who received at least one dose of study drug (RP103) with at least one post-baseline NPMDS assessment and an evaluable Week 24 NPMDS assessment within the protocol specified window.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 18
units on a scale
  Section I | -0.3 (0.7)
  Section II | 0.1 (1.1)
  Section III | -0.6 (1.2)
  Section IV | 0.0 (4.0)
Statistical Analysis 1: Comparison: Cysteamine Bitartrate Delayed-release; Section I - Current Function Null hypothesis = change from baseline is 0; Test type: Other; p = 0.1875, Wilcoxon Signed Rank
Statistical Analysis 2: Comparison: Cysteamine Bitartrate Delayed-release; Section II - System Specific Involvement Null hypothesis = change from baseline is 0; Test type: Other; p = 1.0000, Wilcoxin Signed Rank
Statistical Analysis 3: Comparison: Cysteamine Bitartrate Delayed-release; Section III - Current Clinical Assessment Null hypothesis = change from baseline is 0; Test type: Other; p = 0.0781, Wilcoxin Signed Rank
Statistical Analysis 4: Comparison: Cysteamine Bitartrate Delayed-release; Section IV - Quality of Life Null hypothesis = change from baseline is 0; Test type: Other; p = 0.2941, t-test, 2 sided; One-sample t-test

2. Secondary Outcome: Change From Baseline in Glutathione
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24
Population: The pharmacodynamic (PD) analysis set included all participants who received at least one dose of study drug and had at least one post-baseline PD assessment. Participants with available data at each time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 26
µmol/L
  Week 4: number analyzed (Participants) | 20
  Week 4 | 16.8 (277.1)
  Week 8: number analyzed (Participants) | 21
  Week 8 | 141.5 (275.5)
  Week 12: number analyzed (Participants) | 23
  Week 12 | 10.2 (419.4)
  Week 16: number analyzed (Participants) | 19
  Week 16 | 88.7 (343.9)
  Week 20: number analyzed (Participants) | 17
  Week 20 | 51.4 (207.8)
  Week 24: number analyzed (Participants) | 18
  Week 24 | 122.4 (244.8)

3. Secondary Outcome: Change From Baseline in Glutathione Disulfide
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24
Population: PD analysis set participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 26
µmol/L
  Week 4: number analyzed (Participants) | 20
  Week 4 | 29.4 (96.8)
  Week 8: number analyzed (Participants) | 21
  Week 8 | -9.8 (43.9)
  Week 12: number analyzed (Participants) | 23
  Week 12 | 18.8 (105.3)
  Week 16: number analyzed (Participants) | 19
  Week 16 | -11.2 (46.2)
  Week 20: number analyzed (Participants) | 17
  Week 20 | 0.8 (7.1)
  Week 24: number analyzed (Participants) | 18
  Week 24 | -11.5 (47.6)

4. Secondary Outcome: Change From Baseline in Lactic Acid
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24
Population: PD analysis set participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 31
mmol/L
  Week 4: number analyzed (Participants) | 28
  Week 4 | 0.2 (1.0)
  Week 8: number analyzed (Participants) | 25
  Week 8 | 0.4 (1.6)
  Week 12: number analyzed (Participants) | 27
  Week 12 | 0.3 (2.4)
  Week 16: number analyzed (Participants) | 26
  Week 16 | 0.1 (1.2)
  Week 20: number analyzed (Participants) | 24
  Week 20 | 0.1 (1.1)
  Week 24: number analyzed (Participants) | 27
  Week 24 | 0.0 (1.2)

5. Secondary Outcome: Change From Baseline in 6 Minute Walk Test
Description: The investigator selected the two most preeminent symptoms for each participant during the screening visit from the following: Myopathy, dystonia, ataxia, retarded motor development, reduced activities of daily living, and vision. The 2 symptoms selected for each participant were then assessed at each subsequent study visit.
  Myopathy was assessed using the 6 minute walk test, which measures the distance walked in a 6 minute walk test.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24
Population: Participants who received at least one dose of study drug (RP103) and had at least one post-baseline 6 minute walk test assessment and for whom myopathy was prespecified as a preeminent symptom and with available data at each time point.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 15
meters
  Week 4: number analyzed (Participants) | 13
  Week 4 | -23.5 (86.3)
  Week 8: number analyzed (Participants) | 11
  Week 8 | -36.2 (73.3)
  Week 12: number analyzed (Participants) | 10
  Week 12 | -14.5 (71.5)
  Week 16: number analyzed (Participants) | 10
  Week 16 | -21.3 (90.6)
  Week 20: number analyzed (Participants) | 9
  Week 20 | 21.3 (61.9)
  Week 24: number analyzed (Participants) | 9
  Week 24 | -18.9 (123.9)

6. Secondary Outcome: Change From Baseline in Jamar Dynamometer Hand Strength
Description: The investigator selected the two most preeminent symptoms for each participant during the screening visit from the following: myopathy, dystonia, ataxia, retarded motor development, reduced activities of daily living, and vision. The 2 symptoms selected for each participant were then assessed at each subsequent study visit.
  Myopathy was assessed using standard grip strength evaluation, which measures hand strength in both hands using a Jamar dynamometer.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24
Population: Participants who received at least one dose of study drug (RP103) and had at least one post-baseline Jamar hand strength assessment and for whom myopathy was prespecified as a preeminent symptom and with available data at each time point.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 9
kg
  Week 4 - Left hand | 1.3 (2.4)
  Week 8 - Left hand: number analyzed (Participants) | 8
  Week 8 - Left hand | 1.1 (2.3)
  Week 12 - Left hand: number analyzed (Participants) | 7
  Week 12 - Left hand | 1.3 (2.6)
  Week 16 - Left hand: number analyzed (Participants) | 7
  Week 16 - Left hand | 0.0 (3.3)
  Week 20 - Left hand: number analyzed (Participants) | 7
  Week 20 - Left hand | 0.7 (3.1)
  Week 24 - Left hand: number analyzed (Participants) | 6
  Week 24 - Left hand | 1.3 (2.2)
  Week 4 - Right hand | 0.5 (3.0)
  Week 8 - Right hand: number analyzed (Participants) | 8
  Week 8 - Right hand | 1.6 (2.1)
  Week 12 - Right hand: number analyzed (Participants) | 7
  Week 12 - Right hand | 1.6 (2.6)
  Week 16 - Right hand: number analyzed (Participants) | 7
  Week 16 - Right hand | 0.7 (2.9)
  Week 20 - Right hand: number analyzed (Participants) | 7
  Week 20 - Right hand | 0.9 (2.4)
  Week 24 - Right hand: number analyzed (Participants) | 6
  Week 24 - Right hand | 1.2 (2.1)

7. Secondary Outcome: Change From Baseline in Barry-Albright Dystonia Scale Total Score
Description: The investigator selected the two most preeminent symptoms for each participant during the screening visit from the following: myopathy, dystonia, ataxia, retarded motor development, reduced activities of daily living, and vision. The 2 symptoms selected for each participant were then assessed at each subsequent study visit.
  Dystonia symptoms were assessed using the Barry-Albright Dystonia Scale for Dystonia. Participants were assessed for dystonia in each of the following regions: eyes, mouth, neck, trunk, and each upper and lower extremity (8 body regions) on a scale from 0 (absent) to 4 (severe symptoms). The individual scores were summed to calculate the total score which ranges from 0 (dystonia absent) to 32 (severe dystonia).
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24
Population: Participants who received at least one dose of study drug (RP103) and had at least one post-baseline dystonia assessment and for whom dystonia was prespecified as a preeminent symptom and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 4
units on a scale
  Week 4 | 1.3 (1.0)
  Week 8: number analyzed (Participants) | 3
  Week 8 | 0.7 (0.6)
  Week 12: number analyzed (Participants) | 3
  Week 12 | 0.3 (3.1)
  Week 16: number analyzed (Participants) | 3
  Week 16 | 0.3 (3.1)
  Week 20: number analyzed (Participants) | 3
  Week 20 | -0.7 (4.7)
  Week 24: number analyzed (Participants) | 3
  Week 24 | 0.7 (3.5)

8. Secondary Outcome: Change From Baseline in Friedreich Ataxia Rating Scale
Description: The investigator selected the two most preeminent symptoms for each participant during the screening visit from the following: myopathy, dystonia, ataxia, retarded motor development, reduced activities of daily living, and vision. The 2 symptoms selected for each participant were then assessed at each subsequent study visit.
  Ataxia was assessed using the Friedreich Ataxia Rating Scale (FARS). FARS comprises a functional ataxia staging score of overall mobility (score 0 to 6), an assessment of the activities of daily living (ADL) (score 0 to 36) and a neurological assessment (score from 0 to 117) which is composed of bulbar (score 0-11), upper limb (score 0- 36) and lower limb (score 0-16), peripheral nerve (score 0-26) and upright stability/gait (score 0-28). The scores were summed to calculate the total score which ranges from 0 to 159. A higher score indicates a greater level of disability.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24
Population: Participants who received at least one dose of study drug (RP103) and had at least one post-baseline ataxia assessment and for whom ataxia was prespecified as a preeminent symptom and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 4
units on a scale
  Week 4 | 16.9 (27.2)
  Week 8 | 13.9 (25.6)
  Week 12 | 15.9 (23.1)
  Week 16 | 19.4 (23.0)
  Week 20 | 16.5 (21.5)
  Week 24 | 20.5 (18.5)

9. Secondary Outcome: Change From Baseline in Gross Motor Function
Description: The investigator selected the two most preeminent symptoms for each participant during the screening visit from the following: myopathy, dystonia, ataxia, retarded motor development, reduced activities of daily living, and vision. The 2 symptoms selected for each participant were then assessed at each subsequent study visit.
  Retarded motor development was assessed using the Gross Motor Function Measure (GMFM)-88 which consists of 88 items scored on a scale of 0 to 3:
  0: Does not initiate the task;
  1. Initiates the task (completes < 10%);
  2. Partially completes the task (10 to 99%);
  3. Completes the task (100%).
  The 88 items are grouped into five dimensions: 1) lying and rolling, 2) sitting, 3) crawling and kneeling, 4) standing, and 5) walking, running and jumping. Scores are expressed as a percentage of the maximum score for that dimension. The total score is the average of the 5 the percentage scores where higher scores indicate better performance.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24
Population: Participants who received at least one dose of study drug (RP103) and had at least one post-baseline gross motor function assessment and for whom retarded motor development was prespecified as a preeminent symptom and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 12
units on a scale
  Week 4 | 0.4 (4.3)
  Week 8 | 0.9 (7.9)
  Week 12 | 0.5 (3.6)
  Week 16 | 4.4 (5.6)
  Week 20 | 4.0 (8.2)
  Week 24 | 2.2 (8.2)

10. Secondary Outcome: Change From Baseline in Modified Lansky Play Performance Scale
Description: The investigator selected the 2 most preeminent symptoms for each participant during the screening visit from the following: myopathy, dystonia, ataxia, retarded motor development, reduced activities of daily living, and vision. The 2 symptoms were assessed at each subsequent study visit.
  Reduced activities of daily living was assessed using the modified Lansky Play Performance Scale, completed by parents based on their child's activity in the past week, where 100=fully active; 90=minor restrictions in strenuous physical activity; 80=active, gets tired more quickly; 70=greater restriction of play, less time spent in play activity; 60=up and around, active play minimal; quieter activities; 50=lying around much of the day; no active playing, all quiet play and activities; 40=mainly in bed; quiet activities; 30=bedbound; needs assistance even for quiet play; 20=sleeps often; play limited to very passive activities; 10=doesn't play or get out of bed; 5=unresponsive 0=dead
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24
Population: Participants who received at least one dose of study drug (RP103) and had at least one post-baseline Lansky play performance scale assessment and for whom reduced activities of daily living was prespecified as a preeminent symptom and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cysteamine Bitartrate Delayed-release
Number analyzed (Participants) | 6
units on a scale
  Week 4: number analyzed (Participants) | 5
  Week 4 | -2.0 (4.5)
  Week 8: number analyzed (Participants) | 5
  Week 8 | -6.0 (8.9)
  Week 12: number analyzed (Participants) | 5
  Week 12 | -2.0 (4.5)
  Week 16: number analyzed (Participants) | 5
  Week 16 | 2.0 (11.0)
  Week 20: number analyzed (Participants) | 5
  Week 20 | -4.0 (11.4)
  Week 24: number analyzed (Participants) | 5
  Week 24 | -6.0 (8.9)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Cysteamine Bitartrate Delayed-release
All-Cause Mortality (participants affected / at risk) | 1/36
Serious Adverse Events (participants affected / at risk) | 11/36
Other Adverse Events (participants affected / at risk) | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cysteamine Bitartrate Delayed-release (N=36)
Atrioventricular block complete (Cardiac disorders) | 1
Atrioventricular block second degree (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Adenovirus infection (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Convulsion (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cysteamine Bitartrate Delayed-release (N=36)
Sinus tachycardia (Cardiac disorders) | 1
Motion sickness (Ear and labyrinth disorders) | 1
Eye movement disorder (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 2
Mydriasis (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 4
Breath odour (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 15
Eructation (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 12
Retching (Gastrointestinal disorders) | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 21
Asthenia (General disorders) | 1
Chest pain (General disorders) | 2
Fatigue (General disorders) | 11
Gait disturbance (General disorders) | 2
Malaise (General disorders) | 1
Pyrexia (General disorders) | 12
Bursitis infective (Infections and infestations) | 1
Croup infectious (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Influenza (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 4
Oral herpes (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 3
Rhinovirus infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Viral infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Foot fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 2
Radial head dislocation (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bicarbonate decreased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Clostridium test positive (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Respiratory rate decreased (Investigations) | 1
Weight decreased (Investigations) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 14
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Posture abnormal (Musculoskeletal and connective tissue disorders) | 1
Akathisia (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 4
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dystonia (Nervous system disorders) | 3
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 7
Lethargy (Nervous system disorders) | 8
Migraine (Nervous system disorders) | 1
Parkinsonian rest tremor (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Speech disorder (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 3
Abnormal behaviour (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 2
Mental status changes (Psychiatric disorders) | 1
Mood swings (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Tic (Psychiatric disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 1
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 7
Pallor (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any Investigator/institution that plans on presenting or publishing results provide written notification of their request a minimum of 60 days prior to presentation or publication. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsors' Intellectual Property rights .